CLINICAL TRIAL: NCT05453084
Title: Evaluation of the Effectiveness of a Physical Exercise Intervention on Quality of Life and Symptom Profile of Patients With Irritable Bowel Syndrome (IBS).
Brief Title: Exercise and Irritable Bowel Syndrome (IBS)
Acronym: AF_IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Alberto R Osella, Principal Investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSDebellis
Record Dates: First submitted 2022-06-09; First posted 2022-07-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-12

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome; Exercise; Gastrointestinal Function; Physical activity
MeSH Terms: conditions — Irritable Bowel Syndrome; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): The exercise intervention tool will be Fitwalking, which is structured, organized, supervised and administered through a "Walking Group"
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — The intervention includes an individualized exercise program in terms of Frequency, Intensity, Time, Type, Volume and Progression (FITT-VP).

SUMMARY:
Specific Aim 1: As shown in the literature, exercise can be a useful tool for treating and improving functional GI disorders. Therefore, the aim is to estimate the effectiveness of an exercise intervention on IBS symptoms as measured by a reduction of at least 50 score points on the IBS- Symptom Severity Scale (IBS-SSS) questionnaire.

DETAILED DESCRIPTION:
Inclusion criteria:

Adult patients (18-65 years old) referred to the "Outpatient Clinic for Celiac Disease and Functional Disorders" who met the Rome III-IV criteria for IBS-D and were referred by their local General Practitioner.

Exclusion criteria:

Presence of severe heart, liver, neurological or psychiatric disease or GI disease other than IBS (e.g., inflammatory bowel disease, celiac disease) that could explain the current symptoms.

Patients who have previously followed a diet low in particular substances (e.g., low fermentable oligosaccharides, disaccharides, monosaccharides, and polyols - FODMAP -) diet, vegan diet, a gluten-free diet).

Antidepressant use All patients will receive detailed verbal and written information about the study before giving their written consent.

Methodology: V1. (Screening). Patients will be informed about the objective of the study; V2. (Day 0). Seven days after the screening visit, patients will return for the outpatient visit. At this time, patients will complete the symptom questionnaires. During this visit, blood and biological samples (urine, feces) will be taken; anthropometrical measurements and bioimpedance analysis (BIA) will be carried out. Additionally, ECG will be performed at the Cardiology Unit. V3. (pre-treatment). Seven days before the start of the exercise intervention, the enrolled subjects, only after submitting the certificate of physical fitness issued by their doctor or general practitioner (GP), will undergo three field physical tests for the initial assessment of their fitness. V4. (treatment). Treatment begins after assessing the baseline level of physical activity through analysis of the results of the three field tests. V5. (post-treatment). In the seven days following the end of the Physical Exercise intervention, the subjects are assessed again using the three field tests. V6. (Day 90).

End of treatment visit. During this visit, completed questionnaires will be collected, including the symptom diary and daily exercise diary; in addition, patients will complete the symptom questionnaires (IBS-SSS and GSRS). An anthropometric and bioimpedance analysis will also be performed, and potential adverse events during the intervention period will be assessed. Blood and biological samples necessary for the instrumental evaluations in the study will be taken.

Physical Exercise Intervention: The exercise intervention tool will be Fitwalking, which is structured, organized, supervised, and administered through a "Walking Group". Fitwalking is a motor-sport activity that has innumerable potential for health and physical well-being. Fitwalking is a type of training based on walking, carried out with a precise technique, which allows you to walk well and be faster, thus producing positive metabolic effects and improving physical efficiency. Fitwalking is an aerobic activity of moderate intensity in which the workload produces progressive adaptations and allows for improved recovery and load increase over time. An effective prescription includes a systematically designed and individualized exercise program in terms of Frequency, Intensity, Time, Type, Volume, and Progression (FITT-VP). These parameters are briefly described below:

Frequency. Exercise (walking) will be carried out outdoors on an urban route 3 times a week, on non-consecutive days, for 12 weeks.

Intensity. The intensity of the exercise (50/75% of HRmax) will be monitored through the use of the heart rate monitor and will be personalized through the Tanaka formula. In addition, to measure pace we will use the TALK TEST (a standardized and validated survey tool based on the ability of the exercising subject to holding a conversation), and to measure the perception of fatigue we will use the modified BORG scale (on a scale of 0-10, a perception of 5-6 is needed).

Type. The type of exercise is moderate aerobic with a speed ranging from 5 to 10 km/h. The single outing lasting 60' will be structured as follows:

* Warm-up: 5'
* Normal walk: 10'
* Sustained walking: 30'
* Fast walking: 10'
* Cool-down: 5' Time. Each walk will be led by a walking leader (Master's Degree in Science and Techniques of Preventive and Adapted Motor Activities).

Volume. Participants in the project will perform 180' minutes per week of aerobic exercise of moderate intensity, through walking in groups as per the ACSM (The American College of Sports Medicine) guidance on preventive health. However, participants may also increase their exercise volume through other activities outside the project. All exercise data, both within and outside the project, will be recorded in a daily diary for the assessment of energy expenditure (see appendix).

Progression. The FITT components (Frequency, Intensity, Type, and Time) can be modified and increased according to the subjects' abilities and improvements, to achieve the recommended volume of exercise as per the ACSM (The American College of Sports Medicine) guidance on preventive health.

Statistical analysis. This study aims to evaluate the effectiveness of exercise in symptom management of patients with IBS compared to standard dietary advice. The collected data will be grouped and summarized concerning demographic variables, baseline characteristics, and efficacy and safety assessments. Exploratory analyses will be performed using descriptive statistics. Data will be presented (as mean - standard deviation - SD, unless otherwise stated) for both the intention-to-treat population (i.e., all patients who exercised) and the per-protocol population (i.e., all patients who completed the study without major protocol violations). Patients who discontinued the study will also be listed, and their reasons described analytically. Categorical variables will be compared with the X2 test. Two-tailed p-values <0.05 will be considered statistically significant.

Statistical analysis will be performed using the Generalized Estimating Equation procedure to estimate the effect of interventions on the outcome (IBS-SSS). These models are instrumental in biomedical studies to evaluate the change in outcome in the presence of covariates. To overcome the non-normal distribution, a gamma distribution of the outcome will be assumed, and the identity link will be used. The structure of the covariance between the different measurements will be explored with special programs. The results will be expressed in the natural scale of the outcome measurement as the mean and the corresponding 95% confidence intervals. Marginal effects of interventions will also be estimated for different covariates or combinations of covariates. All statistical analyses will be performed using the statistical software Stata 17 (StataCorp, 4905 Lakeway Drive, College Station, Texas 77845 USA). In particular, the -xtgee- command will be used, and the statistical structure of the covariance will be explored with the -qic- command.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred to the "Outpatient Clinic for Celiac Disease and Functional Disorders" who meet the Rome III-IV criteria for IBS-D and referred by their local General Practitioner.

Exclusion Criteria:

* Presence of severe heart, liver, neurological or psychiatric disease or GI disease other than IBS (e.g., inflammatory bowel disease, celiac disease) that could explain the current symptoms.

Patients who have previously followed a diet low in particular substances (e.g., low FODMAPs, vegan diet, gluten-free diet).

Antidepressant use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Symptom assessment | Baseline and after 3 months
  To evaluate the effectiveness of an exercise intervention on IBS symptoms as measured by a change in the IBS-Symptom Severity Scale (IBS-SSS) questionnaire score from baseline.
  The IBS-SSS is a validated questionnaire for gastrointestinal symptoms and provides a global measure of symptom severity by assessing five items ("severity of abdominal pain", "frequency of abdominal pain", "severity of abdominal distension", "dissatisfaction with bowel habits", "impact of symptoms on quality of life") on a visual analogue scale. The values of the five items are added together to give a total score between 0 and 500. Cases are then classified as 'mild' (75 to 175), 'moderate' (175 to 300) and 'severe' (>300).

SECONDARY OUTCOMES:
Gatroduodenal permeability | Baseline and after 3 months
  will be assessed by administering a mixture of sucrose-lactulose-mannitol-sucralose and measuring their gastrointestinal absorption by urinary excretion of these sugars.
Evaluation of Barrier peptide integrity | Baseline and after 3 months
  Zonulin, I-FABP and DAO and D-lactate assays will be performed using commercially available ELISAs
Intestinal microbiota analysis | Baseline and after 3 months
  Evaluation of any differences in the intestinal microbial population in the different disease patterns considered will be performed using appropriate genetic and molecular investigations (Illumina/Solexa Genetic Analyzer HiSeq) on the patients' stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Alberto R Osella, PhD, Principal Investigator — National Institute for Digestive Diseases IRCCS " Saverio de Bellis"
Locations (1):
- Laboratory of Epidemiology and Statistic- IRCCS De Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orlando A, Tutino V, Notarnicola M, Riezzo G, Linsalata M, Clemente C, Prospero L, Martulli M, D'Attoma B, De Nunzio V, Russo F. Improved Symptom Profiles and Minimal Inflammation in IBS-D Patients Undergoing a Long-Term Low-FODMAP Diet: A Lipidomic Perspective. Nutrients. 2020 Jun 2;12(6):1652. doi: 10.3390/nu12061652. PMID 32498383
- [Background] Johannesson E, Jakobsson Ung E, Sadik R, Ringstrom G. Experiences of the effects of physical activity in persons with irritable bowel syndrome (IBS): a qualitative content analysis. Scand J Gastroenterol. 2018 Oct-Nov;53(10-11):1194-1200. doi: 10.1080/00365521.2018.1519596. Epub 2018 Nov 25. PMID 30472905
- [Background] Johannesson E, Simren M, Strid H, Bajor A, Sadik R. Physical activity improves symptoms in irritable bowel syndrome: a randomized controlled trial. Am J Gastroenterol. 2011 May;106(5):915-22. doi: 10.1038/ajg.2010.480. Epub 2011 Jan 4. PMID 21206488
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Prospero L, Riezzo G, Linsalata M, Orlando A, D'Attoma B, Russo F. Psychological and Gastrointestinal Symptoms of Patients with Irritable Bowel Syndrome Undergoing a Low-FODMAP Diet: The Role of the Intestinal Barrier. Nutrients. 2021 Jul 19;13(7):2469. doi: 10.3390/nu13072469. PMID 34371976
- [Background] Linsalata M, Riezzo G, Orlando A, D'Attoma B, Prospero L, Tutino V, Notarnicola M, Russo F. The Relationship between Low Serum Vitamin D Levels and Altered Intestinal Barrier Function in Patients with IBS Diarrhoea Undergoing a Long-Term Low-FODMAP Diet: Novel Observations from a Clinical Trial. Nutrients. 2021 Mar 21;13(3):1011. doi: 10.3390/nu13031011. PMID 33801020
- [Background] Franco I, Bianco A, Diaz MDP, Bonfiglio C, Chiloiro M, Pou SA, Becaria Coquet J, Mirizzi A, Nitti A, Campanella A, Leone CM, Caruso MG, Correale M, Osella AR. Effectiveness of two physical activity programs on non-alcoholic fatty liver disease. a randomized controlled clinical trial. Rev Fac Cien Med Univ Nac Cordoba. 2019 Feb 27;76(1):26-36. doi: 10.31053/1853.0605.v76.n1.21638. PMID 30882339
- [Background] Notarnicola M, Caruso MG, Tutino V, Bonfiglio C, Cozzolongo R, Giannuzzi V, De Nunzio V, De Leonardis G, Abbrescia DI, Franco I, Intini V, Mirizzi A, Osella AR. Significant decrease of saturation index in erythrocytes membrane from subjects with non-alcoholic fatty liver disease (NAFLD). Lipids Health Dis. 2017 Aug 23;16(1):160. doi: 10.1186/s12944-017-0552-0. PMID 28830448
- [Background] Tutino V, De Nunzio V, Caruso MG, Bonfiglio C, Franco I, Mirizzi A, De Leonardis G, Cozzolongo R, Giannuzzi V, Giannelli G, Notarnicola M, Osella AR. Aerobic Physical Activity and a Low Glycemic Diet Reduce the AA/EPA Ratio in Red Blood Cell Membranes of Patients with NAFLD. Nutrients. 2018 Sep 13;10(9):1299. doi: 10.3390/nu10091299. PMID 30217048
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Background] Riegler G, Esposito I. Bristol scale stool form. A still valid help in medical practice and clinical research. Tech Coloproctol. 2001 Dec;5(3):163-4. doi: 10.1007/s101510100019. PMID 11875684
- [Background] Hanson S, Jones A. Is there evidence that walking groups have health benefits? A systematic review and meta-analysis. Br J Sports Med. 2015 Jun;49(11):710-5. doi: 10.1136/bjsports-2014-094157. Epub 2015 Jan 19. PMID 25601182
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] Foster C, Porcari JP, Anderson J, Paulson M, Smaczny D, Webber H, Doberstein ST, Udermann B. The talk test as a marker of exercise training intensity. J Cardiopulm Rehabil Prev. 2008 Jan-Feb;28(1):24-30; quiz 31-2. doi: 10.1097/01.HCR.0000311504.41775.78. PMID 18277826
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Pengpid S, Peltzer K. Sedentary Behaviour, Physical Activity and Life Satisfaction, Happiness and Perceived Health Status in University Students from 24 Countries. Int J Environ Res Public Health. 2019 Jun 13;16(12):2084. doi: 10.3390/ijerph16122084. PMID 31200427
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Laukkanen R, Oja P, Pasanen M, Vuori I. Validity of a two kilometre walking test for estimating maximal aerobic power in overweight adults. Int J Obes Relat Metab Disord. 1992 Apr;16(4):263-8. PMID 1318280
- [Background] Pearn J, Bullock K. A portable hand-grip dynamometer. Aust Paediatr J. 1979 Jun;15(2):107-9. doi: 10.1111/j.1440-1754.1979.tb01200.x. No abstract available. PMID 485989
- [Background] Ulijaszek SJ, Kerr DA. Anthropometric measurement error and the assessment of nutritional status. Br J Nutr. 1999 Sep;82(3):165-77. doi: 10.1017/s0007114599001348. PMID 10655963
- [Background] Hoeger WW, Hopkins DR. A comparison of the sit and reach and the modified sit and reach in the measurement of flexibility in women. Res Q Exerc Sport. 1992 Jun;63(2):191-5. doi: 10.1080/02701367.1992.10607580. No abstract available. PMID 1585066
- [Background] Khalil SF, Mohktar MS, Ibrahim F. The theory and fundamentals of bioimpedance analysis in clinical status monitoring and diagnosis of diseases. Sensors (Basel). 2014 Jun 19;14(6):10895-928. doi: 10.3390/s140610895. PMID 24949644
- [Background] Midenfjord I, Polster A, Sjovall H, Tornblom H, Simren M. Anxiety and depression in irritable bowel syndrome: Exploring the interaction with other symptoms and pathophysiology using multivariate analyses. Neurogastroenterol Motil. 2019 Aug;31(8):e13619. doi: 10.1111/nmo.13619. Epub 2019 May 5. PMID 31056802
- [Background] Garner DM, Garfinkel PE. The Eating Attitudes Test: an index of the symptoms of anorexia nervosa. Psychol Med. 1979 May;9(2):273-9. doi: 10.1017/s0033291700030762. PMID 472072
- [Background] Bertolotti G, Zotti AM, Michielin P, Vidotto G, Sanavio E. A computerized approach to cognitive behavioural assessment: an introduction to CBA-2.0 primary scales. J Behav Ther Exp Psychiatry. 1990 Mar;21(1):21-7. doi: 10.1016/0005-7916(90)90045-m. PMID 2197296
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928
- [Background] ZUNG WW. A SELF-RATING DEPRESSION SCALE. Arch Gen Psychiatry. 1965 Jan;12:63-70. doi: 10.1001/archpsyc.1965.01720310065008. No abstract available. PMID 14221692
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] The psychological results of 438 patients with persisting GERD symptoms by Symptom Checklist 90-Revised (SCL-90-R) questionnaire: Retraction. Medicine (Baltimore). 2018 Jun;97(22):e10768. doi: 10.1097/MD.0000000000010768. No abstract available. PMID 29851782
- [Background] Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998 Feb;43(2):400-11. doi: 10.1023/a:1018831127942. PMID 9512138
- [Background] Linsalata M, Riezzo G, D'Attoma B, Clemente C, Orlando A, Russo F. Noninvasive biomarkers of gut barrier function identify two subtypes of patients suffering from diarrhoea predominant-IBS: a case-control study. BMC Gastroenterol. 2018 Nov 6;18(1):167. doi: 10.1186/s12876-018-0888-6. PMID 30400824
- [Background] Kataoka K. The intestinal microbiota and its role in human health and disease. J Med Invest. 2016;63(1-2):27-37. doi: 10.2152/jmi.63.27. PMID 27040049
- [Background] Garcia Regueiro JA, Rius MA. Rapid determination of skatole and indole in pig back fat by normal-phase liquid chromatography. J Chromatogr A. 1998 Jun 5;809(1-2):246-51. doi: 10.1016/s0021-9673(98)00191-5. PMID 9677718
- [Result] Simren M, Tack J. New treatments and therapeutic targets for IBS and other functional bowel disorders. Nat Rev Gastroenterol Hepatol. 2018 Oct;15(10):589-605. doi: 10.1038/s41575-018-0034-5. PMID 29930260
- [Derived] Prospero L, Riezzo G, D'Attoma B, Ignazzi A, Bianco A, Franco I, Curci R, Campanella A, Bagnato CB, Porcelli P, Giannelli G, Russo F. The impact of locus of control on somatic and psychological profiles of patients with irritable bowel syndrome engaging in aerobic exercise. Sci Rep. 2025 Feb 1;15(1):3966. doi: 10.1038/s41598-025-88466-7. PMID 39893252